CLINICAL TRIAL: NCT02148939
Title: Dipyrone Nullifies Aspirin Antiplatelet Effects in Stroke-Patients
Brief Title: Antiplatelet Effects in Stroke-Patients
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Division of Cardiology, Pulmonary Diseases, Vascular Medicine, Heinrich-Heine University, Duesseldorf
Other Study IDs: Stroke
Record Dates: First submitted 2014-05-16; First posted 2014-05-29 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; Antiplatelet Effects; aspirin; metamizole; dipyrone
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Many patients suffer from acute and chronic pain. The incidence of chronic pain correlates with increased age. Most of patients rely on analgesic medication to control the pain. Dipyrone is an extensively used drug in Western and Eastern Europe as well as Central and South America, largely due to its favorable analgesic and antipyretic effects in conjunction with a low incidence of gastrointestinal complications when compared to other non-steroidal anti-inflammatory drugs (NSAIDs).

Aspirin is the backbone of antiplatelet therapy in patients after ischemic stroke. However, it is known that there are substantial inter-individual response variabilities to antiplatelet medication. Furthermore, patients with impaired response to aspirin have a significant higher risk of recurrent cerebrovascular events. The investigators have recently shown that co-medication with aspirin and dipyrone in patients with coronary artery disease lead to insufficient antiplatelet effects of aspirin.

The incidence of chronic pain is very high in patients with ischemic stroke. Therefore, in this study the investigators aim to examine, if co-medication of aspirin and dipyrone interaction also occurs in patients after ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with ischemic stroke and ASS-medication (80-320 mg/day) with/without analgesic comedication

Exclusion Criteria:

* Reanimation
* cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Laboratory response to aspirin therapy in metamizole co-medicated Stroke patients | Baseline

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE Events) during hospital stay | participants are followed until discharge up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amin Polzin, MD, Principal Investigator — Klinik für Kardiologie, Pneumologie und Angiologie, Universtiätsklinikum Düsseldorf; Tobias Zeus, MD, Study Chair — Klinik für Kardiologie, Pneumologie und Angiologie, Universtiätsklinikum Düsseldorf
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

REFERENCES:
- [Derived] Dannenberg L, Erschoff V, Bonner F, Gliem M, Jander S, Levkau B, Kelm M, Hohlfeld T, Zeus T, Polzin A. Dipyrone comedication in aspirin treated stroke patients impairs outcome. Vascul Pharmacol. 2016 Dec;87:66-69. doi: 10.1016/j.vph.2016.06.003. Epub 2016 Jun 11. PMID 27301652
- See also: Related Info — http://www.uniklinik-duesseldorf.de/kardiologie